CLINICAL TRIAL: NCT03375151
Title: An Examination of the Use of Electrophysiological Brain Monitoring to Direct the Treatment of Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brainmarc Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLD13
Record Dates: First submitted 2017-12-13; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EEG based feedback (Experimental): The therapist will give feedback to the participants during the exercise based on their performance.and use the feedback from the EEG analyzed data to direct cognitive therapy based on the therapist's guidance to maximize the intensity and duration of the patient's high brain engagement Index (BEI) during exercise.
  Interventions: Device: EEG based feedback; Behavioral: Standard practice based feedback
- Standard practice based feedback (Other): The therapist will give feedback to the participants during the exercise based on their performance.
  Interventions: Behavioral: Standard practice based feedback
- No feedback (Other): The participants will perform the exercise without feedback during practice.
  Interventions: Behavioral: No feedback

INTERVENTIONS:
Device: EEG based feedback — Participants will participate in cognitive training sessions. The therapist will use feedback from the EEG analyzed data to direct the cognitive therapy based on the therapist's guidance to maximize the intensity and duration of the patient's high brain engagement Index (BEI) during exercise.
  Arms: EEG based feedback
Behavioral: Standard practice based feedback — Participants will participate in cognitive training sessions. The therapist will give feedback to the participants during the exercise based on their performance only according to the his therapist standard practice.
  Arms: EEG based feedback; Standard practice based feedback
Behavioral: No feedback — Participants will participate in cognitive training sessions. The therapist will not guide them during the sessions.
  Arms: No feedback

SUMMARY:
The problem of cognitive decline among the aging population has become a significant health burden, especially in light of the increase in the prevalence of dementia with age For patients with MCI (Mild cognitive impairment) there are various recommendations to deal with the disorder, including behavioral recommendations for physical exercise. Some recommendations could also be found for cognitive practice. However, currently, there is no consensus regarding effective cognitive treatment or practice for MCI. Among the populations suffering from MCI, there is a significant segment of patients with amnestic disorder. For these patients, it seems that cognitive training of memory, including verbal memory, is very important. In recent years, we have developed an effective tool for managing rehabilitation practice by monitoring the patient's engagement with an easy-to-use EEG (electroencephalogram) tool. We have shown in a variety of rehabilitation settings, that when the patient is recruited, the clinical improvement is significantly better. The aim of this study is to evaluate the ability to harness the EEG monitoring of brain engagement to achieve functional improvement in verbal memory training in patients with Amnestic MCI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female above the age of 65 years
* Ability to read, write and understand the Hebrew language so to comply with study demands.
* Diagnosed with Amnestic MCI. Mini Mental State Examination (MMSE), A score of MSSE ≥27 for college educated subjects and MSSE ≥ 26 for all others; and (CDR) Clinical Dementia Rating, 0.5 ≥ CDR
* Diagnosed with memory impairment, Visual Paired Association = VPA (WMS-R), for subjects of ages 65-70, 16.5 ≥ WMS-R and for subjects of age above 71, 15.5 ≥ WMS-R

Exclusion Criteria:

* Diagnosed with major psychiatric or neurological disorder.
* A user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Cognitive test grade | up to 5 weeks
  The difference in grades in a test for evaluation cognitive abilities in a textual assignment between the beginning and the end of the study.

SECONDARY OUTCOMES:
Rey Auditory-Verbal Learning Test | up to 5 weeks
  The difference in grades of Free And Cued Selective Reminding Test (FCSRT) score between the beginning and the end of the study.
Free And Cued Selective Reminding Test | up to 5 weeks
  The difference in grades of Rey Auditory-Verbal Learning Test (RAVLT) score between the beginning and the end of the study.
Rivermead Behavioral Memory Test | up to 5 weeks
  The difference in grades of Rivermead Behavioral Memory Test (RBMT) score between the beginning and the end of the study.
Clinical Global Impression of Change | up to 5 weeks
  The difference in grades of Clinical Global Impression of Change (CGI-C) score between the beginning and the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: David Dvir, Dr., Principal Investigator — Reuth rehabilitation medical center